CLINICAL TRIAL: NCT04142528
Title: ParkinPal: Patient-Centered PD Ambulatory Monitoring System
Brief Title: Patient-Centered PD Ambulatory Monitoring System
Acronym: ParkinPal
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: NR018128-01; 1R43NR018128-01 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Parkinson's Disease: Smartwatch-based sensor assessment of PD symptoms during standard care
  Interventions: Device: ParkinPal

INTERVENTIONS:
Device: ParkinPal — Wear and periodic recording of motion data during daily wear
  Other Names: KinesiaU motor assessment system

SUMMARY:
This a usability study of a wearable sensor platform that utilizes a smartwatch to periodically record motion data. That data is processed in a connected smartphone and translated into symptom scores for dyskinesia, slowness, and tremor. The research subjects will use the wearable system over the course of five weeks, during which a change in therapy regimen is prescribed by the physician. Research analysis will be focused on patient and clinician experiences with the app and its reports.

ELIGIBILITY:
Inclusion Criteria:

* Existing Patient of Collaborating Physician (David E. Riley, MD)
* Diagnosed With Parkinson's Disease
* Hoehn & Yahr Scale I-III
* Ambulatory and capable of using the ParkinPal system
* Able to understand and follow instructions regarding using the device

Exclusion Criteria:

* Any subject that does not meet the subject selection criteria will be excluded from this study. Children will be excluded from this study due to the fact that they are unlikely to have PD. Subjects that are not capable of functioning independently or are so symptomatic as to compromise their safety will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is people with Parkinson's Disease who are patients of David E. Riley, MD. Therefore most participants will reside in the northeast Ohio area.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Useability | 6 weeks
  Following the study, patients will complete questionnaires on their experience with the wearable system.

SECONDARY OUTCOMES:
Symptom scores | 6 weeks
  The recorded scores will be and timing of medication and exercise diary entries will be examined to measure the effect of therapy and therapy regimen change on symptom scores.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies
Locations (1):
- David E. Riley, MD, Warrensville Heights, Ohio, United States